CLINICAL TRIAL: NCT02750280
Title: A Prospective, Randomized, Controlled, Longitudinal Study Using Repeated Measures Design to Evaluate a Porcine Urinary Bladder-Derived Extracellular Matrix (MatriStem®) in the Management of Diabetic Foot Ulcers
Brief Title: A Longitudinal Study to Evaluate an Extracellular Matrix (MatriStem®) for the Treatment of Diabetic Foot Ulcers
Acronym: M-S-DFU-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Calvary Hospital, Bronx, NY (Other)
Collaborators: Integra LifeSciences Corporation (Industry)
Responsible Party: Principal Investigator, Oscar M. Alvarez, PhD, Director, Center for Curative & palliative Wound Care, Calvary Hospital, Bronx, NY
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CA2014-002
Record Dates: First submitted 2016-04-21; First posted 2016-04-25 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Neuropathic Diabetic Foot Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Urinary Bladder matrix (UBM) (Experimental): UBM covered with silicone foam dressing plus total contact cast
  Interventions: Device: MatriStem® [Urinary Bladder Matrix (UBM)]
- Standard Care (Active Comparator): Silicone foam dressing plus total contact cast
  Interventions: Device: Mepilex® [Silicone foam dressing]

INTERVENTIONS:
Device: MatriStem® [Urinary Bladder Matrix (UBM)] — Porcine derived urinary bladder extracellular matrix
  Other Names: MatriStem
  Arms: Urinary Bladder matrix (UBM)
Device: Mepilex® [Silicone foam dressing] — primary wound dressing
  Other Names: Mepilex
  Arms: Standard Care

SUMMARY:
This ia a prospective controlled longitudinal study to evaluate the effects of MatriStem® plus standard local wound care versus standard local wound care alone in the treatment of diabetic foot ulcers (DFUs), as assessed by incidence of complete wound healing by 16 weeks and ulcer recurrence with a 2 year follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects 18-85 years of age with diabetes mellitus (type 1 or type 2)
2. Subject's foot ulcer is on the plantar surface of the foot.
3. DFU has not healed after more than2 months of SOC treatment administered
4. Subject's ulcer must be Wagner type 1 or 2 (uninfected, extending through the dermis and into subcutaneous tissue or granulating but without exposure of tendon, bone, or joint capsule.
5. Subject's wound is free of necrotic debris (post debridement) and clinical infection, should be comprised of healthy, vascular tissue.
6. Subject's Ankle-Brachial Index (ABI) by Doppler method is ≥ 0.7
7. The subject has adequate circulation to the foot to allow for healing. This must be demonstrated by methods described in section 5.1
8. Subject's diabetes is under control as determined by the Investigator
9. Study subject must be reliable, responsible and able to visit the clinic weekly for the full 16 week period. The subject is willing and able to tolerate TCC. Subject is willing to comply with the monthly follow-up regimen for 32 weeks (8 months) The subject is able to return to the clinic if ulcer recurrence occurs
10. Subject or his/her legal representative has read and signed the Institutional Review Board (IRB) approved Informed Consent form before treatment
11. No active malignancy except non-melanoma skin cancer

Exclusion Criteria:

1. Subject has clinical evidence of gangrene on any part of the affected foot
2. Subject has a Wagner type 3 or greater ulceration
3. The subject's ulcer is due to a non-diabetic etiology, Ulcers of arterial, venous stasis, pressure, radiation, traumatic, rheumatoid, vasculitis, collagen vascular disease, or other non-diabetic etiologies
4. Subject has a known sensitivity to bovine or porcine derived devices
5. Subject has one or more medical condition(s) including renal, hepatic, hematological, neurologic, or immune disease that in the opinion of the Investigator would make the subject an inappropriate candidate for this wound healing study
6. Subject has or has had a malignant disease (other than cutaneous epithelioma) not in remission
7. Subject is receiving oral or parenteral corticosteroids, immunosuppressive or cytotoxic agents, or is anticipated to require such agents during the course of the study
8. Subject has chronic osteomyelitis as determined by high resolution ultrasonography
9. Subject's ulcer is infected or accompanied by active cellulitis as determined by the Investigator
10. Subject has any condition(s) that seriously compromises the subject's ability to complete the study
11. Subject is pregnant or lactating at the time of treatment
12. Subject has received growth factor therapy (e.g. autologous platelet-rich plasma gel, bacaplermin, bilayered cell therapy, dermal substitute, extracellular matrix) within two weeks of enrollment. If Santyl or any other collagenase is used, a subject must have a washout period of 2 weeks before MatriStem® can be applied.
13. Subject is currently receiving or has received radiation or chemotherapy within 3 months of randomization
14. Subject has a history of alcohol or drug abuse
15. Subject allergic to a broad spectrum of primary & secondary dressing materials, including occlusive dressings and the adhesives on such dressings.
16. Subject is currently enrolled or participated within the previous 30 days of enrollment in another device, drug or biological trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Incidence of wound healing | 16 weeks

SECONDARY OUTCOMES:
Incidence of ulcer recurrence | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: oscar Alvarez, PhD, Principal Investigator — Calvary Hospital Director, Center for curative and palliative wound care
Locations (1):
- Calvary Hospital Center for Curative and Palliative Wound Care, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No